CLINICAL TRIAL: NCT01306266
Title: A Randomized, Double-blind, Placebo-controlled, Crossover Trial of Rizatriptan 10 mg Oral Disintegrating Tablet for Treatment of Acute Attacks of Chronic, Blast-induced, Post-traumatic Headache in U.S. Military Troops
Brief Title: Study of Rizatriptan in the Treatment of Acute Attacks of Post-traumatic Headache in U.S. Military Troops
Acronym: Maxalt
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Marianne Spevak, Manger, Office of Regulatory Affairs, Henry M. Jackson Foundation for the Advancement of Military Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MAMC 211004
Record Dates: First submitted 2011-02-25; First posted 2011-03-01 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Chronic Post-traumatic Headache
Keywords: active duty; blast induced; headache
MeSH Terms: conditions — Headache | interventions — rizatriptan; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rizatriptan (Active Comparator): initial treatment with Maxalt-MLT 10 mg followed by treatment with placebo
  Interventions: Drug: Rizatriptan
- Placebo (Placebo Comparator): Initial treatment with placebo followed by treatment with Maxalt-MLT 10 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rizatriptan — initial treatment with Maxalt-MLT 10 mg followed by treatment with placebo. Drug is to be taken at onset of a moderate or severe headache
  Other Names: Maxalt
  Arms: rizatriptan
Drug: Placebo — Initial treatment with placebo followed by treatment with Maxalt-MLT 10 mg at onset of a moderate or severe headache.
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the effectiveness of rizatriptan for treating attacks of chronic post-traumatic headache.

DETAILED DESCRIPTION:
Chronic post-traumatic headaches develop in about one third of soliders who have had head trauma caused by a blast. A wide variety of pain medicines, including rizatriptan, are used to treat these headaches in clinical practice. However, the effectiveness has not been established by clinical research studies.

ELIGIBILITY:
Inclusion Criteria:

1. U.S. Army soldier with history of concussion while deployed to a combat zone. Concussion is defined as head trauma with all of the following:
2. No loss of consciousness or loss of consciousness less than 30 minutes.
3. Glasgow Coma Score 13-15 (if known)
4. Symptoms or signs of concussion.
5. Concussion was secondary to primary, secondary, or tertiary blast injury.
6. Headaches started within 7 days of concussion.
7. Headaches have occurred for more than 3 months but not more than 24 months since the precipitating concussion.
8. Headaches occurred 3 to 14 days per month during each of the previous two months.
9. Headaches are migraine type and possess three or more of the following migraine features:
10. moderate or severe pain
11. throbbing or pulsatile pain
12. unilateral or asymmetric pain
13. pain exacerbated by or interfering with routine physical activity
14. nausea or vomiting
15. photosensitivity and phonosensitivity
16. Headaches last 4 or more hours without treatment.
17. Males 18 to 49 years of age.
18. Migraine Disability Assessment Score (MIDAS) greater than 10 or Headache Impact Test-6 (HIT6) score greater than 60.

    -

Exclusion Criteria:

1. Patients with a history of migraine headaches prior to concussion will be excluded.
2. Prior use of any triptan medication for headache.
3. Use of non-opioid analgesic medications 15 or more days per month for the previous month.
4. Use of opioid medications more than 10 days in the previous month.
5. Alcohol consumption of more than two servings (a serving is 2 oz hard liquor, 5 oz wine, or 12 oz beer) per day or more than 3 servings at one time on a weekly basis.
6. Taking two or more medications from the following medication classes: SSRI, SNRI, or TCA.
7. Headache prophylactic medication is allowed but must remain unchanged during the study period.
8. Patients with depression, defined as a PHQ-9 score greater than 15, will be excluded from study participation.
9. PTSD is NOT an exclusion criterion. PTSD will be defined as a clinical diagnosis by a behavioral health provider or PTSD symptom checklist score of 50 or higher.
10. Systolic BP > 140 or diastolic BP > 90 on repeated measurements.
11. Active use of dihydroergotamine.
12. Known coronary artery disease, prior myocardial infarction, history of stroke or TIA, or liver disease.
13. Subjects who will not be available for study-related follow-up visits will be excluded.
14. Patient has cognitive impairment defined as mini-mental status exam score less than 27.
15. Patients undergoing a medical board for headache, sequelae of TBI, or psychiatric disorders will be excluded.
16. Patients suspected of malingering, exaggerating symptoms, or non-compliance will be excluded from study participation.
17. Patient has hemiplegic migraine or basilar migraine.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Headache Severity | 2 hours
  proportion of subjects who obtain headache relief defined as no pain or mild pain two hours after dosing

SECONDARY OUTCOMES:
24 hour Migraine Quality of Life score | 24 hours
  proportions of subjects achieving complete headache relief at 2 hours, sustained headache relief at 24 hours, 24-hour Migraine Quality of Life score, disability 2 hours after dosing, occurrence of associated symptoms, and side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Jay C Erickson, MD, Principal Investigator — U.S. Army Medical Corp. Madigan Army Medical Center
Locations (1):
- Madigan Army Medical Center - Neurology Clinic, Tacoma, Washington, United States